CLINICAL TRIAL: NCT03524339
Title: Perioperative Administration of Tamsulosin vs Placebo to Prevent Postoperative Urinary Retention in Female Pelvic Reconstructive Surgery
Brief Title: Tamsulosin vs Placebo to Prevent Postoperative Urinary Retention in Female Pelvic Reconstructive Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Graham Chapman, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tamsulosin for POUR
Record Dates: First submitted 2018-04-10; First posted 2018-05-14 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Urinary Retention; Lower Urinary Tract Symptoms; Stress Urinary Incontinence; Pelvic Organ Prolapse
MeSH Terms: conditions — Urinary Retention; Lower Urinary Tract Symptoms; Urinary Incontinence, Stress; Pelvic Organ Prolapse | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- Tamsulosin (Experimental)
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Placebo oral capsule — Tamsulosin or placebo will be given for 3 days prior to surgery and one week after surgery to determine its effects on postoperative urinary retention.
  Arms: Placebo
Drug: Tamsulosin — Tamsulosin or placebo will be given for 3 days prior to surgery and one week after surgery to determine its effects on postoperative urinary retention.
  Arms: Tamsulosin

SUMMARY:
This is a placebo controlled randomized controlled trial of perioperative use of tamsulosin to prevent postoperative urinary retention in female pelvic reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older as well as willing and able to provide informed consent
* Patients must be undergoing a scheduled surgery for pelvic organ prolapse or urinary incontinence
* Standard postoperative plan must include admission to the hospital with foley catheterization overnight the night after surgery, and planned removal of foley catheter and active voiding trial on postoperative day 1.

Exclusion Criteria:

* Patient unable or unwilling to provide informed consent
* Severe allergy to sulfa drugs
* Known allergy to tamsulosin or another alpha antagonist medication
* History of urinary retention
* Planned bladder catheterization greater than 24 hours after surgery
* Current use of alpha antagonist medication for hypertension
* End stage renal or liver disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Chapman, Principal Investigator — University Hospitals Case Western Reserve University
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University Hospitals, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hakvoort RA, Dijkgraaf MG, Burger MP, Emanuel MH, Roovers JP. Predicting short-term urinary retention after vaginal prolapse surgery. Neurourol Urodyn. 2009;28(3):225-8. doi: 10.1002/nau.20636. PMID 19130599
- [Background] Chong C, Kim HS, Suh DH, Jee BC. Risk factors for urinary retention after vaginal hysterectomy for pelvic organ prolapse. Obstet Gynecol Sci. 2016 Mar;59(2):137-43. doi: 10.5468/ogs.2016.59.2.137. Epub 2016 Mar 16. PMID 27004205
- [Background] Espaillat-Rijo L, Siff L, Alas AN, Chadi SA, Zimberg S, Vaish S, Davila GW, Barber M, Hurtado EA. Intraoperative Cystoscopic Evaluation of Ureteral Patency: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1378-1383. doi: 10.1097/AOG.0000000000001750. PMID 27824741
- [Background] FitzGerald MP, Brubaker L. The etiology of urinary retention after surgery for genuine stress incontinence. Neurourol Urodyn. 2001;20(1):13-21. doi: 10.1002/1520-6777(2001)20:13.0.co;2-r. PMID 11135378
- [Background] Reitz A, Haferkamp A, Kyburz T, Knapp PA, Wefer B, Schurch B. The effect of tamsulosin on the resting tone and the contractile behaviour of the female urethra: a functional urodynamic study in healthy women. Eur Urol. 2004 Aug;46(2):235-40; discussion 240. doi: 10.1016/j.eururo.2004.04.009. PMID 15245819
- [Background] Pummangura N, Kochakarn W. Efficacy of tamsulosin in the treatment of lower urinary tract symptoms (LUTS) in women. Asian J Surg. 2007 Apr;30(2):131-7. doi: 10.1016/S1015-9584(09)60146-9. PMID 17475584
- [Background] Zhang HL, Huang ZG, Qiu Y, Cheng X, Zou XQ, Liu TT. Tamsulosin for treatment of lower urinary tract symptoms in women: a systematic review and meta-analysis. Int J Impot Res. 2017 Jul;29(4):148-156. doi: 10.1038/ijir.2017.12. Epub 2017 Apr 20. PMID 28424499
- [Background] Madani AH, Aval HB, Mokhtari G, Nasseh H, Esmaeili S, Shakiba M, Shakiba RS, Seyed Damavand SM. Effectiveness of tamsulosin in prevention of post-operative urinary retention: a randomized double-blind placebo-controlled study. Int Braz J Urol. 2014 Jan-Feb;40(1):30-6. doi: 10.1590/S1677-5538.IBJU.2014.01.05. PMID 24642148
- [Background] Akkoc A, Aydin C, Topaktas R, Kartalmis M, Altin S, Isen K, Metin A. Prophylactic effects of alpha-blockers, Tamsulosin and Alfuzosin, on postoperative urinary retention in male patients undergoing urologic surgery under spinal anaesthesia. Int Braz J Urol. 2016 May-Jun;42(3):578-84. doi: 10.1590/S1677-5538.IBJU.2015.0256. PMID 27286124
- [Background] Poylin V, Curran T, Cataldo T, Nagle D. Perioperative use of tamsulosin significantly decreases rates of urinary retention in men undergoing pelvic surgery. Int J Colorectal Dis. 2015 Sep;30(9):1223-8. doi: 10.1007/s00384-015-2294-7. Epub 2015 Jun 23. PMID 26099320
- [Derived] Chapman GC, Sheyn D, Slopnick EA, Roberts K, El-Nashar SA, Henderson JW, Mangel J, Hijaz AK, Pollard RR, Mahajan ST. Tamsulosin vs placebo to prevent postoperative urinary retention following female pelvic reconstructive surgery: a multicenter randomized controlled trial. Am J Obstet Gynecol. 2021 Sep;225(3):274.e1-274.e11. doi: 10.1016/j.ajog.2021.04.236. Epub 2021 Apr 21. PMID 33894146

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Tamsulosin
Started | 66 | 66
Completed | 57 | 62
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tamsulosin | Total
Number analyzed (Participants) | 57 | 62 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.9) | 61.0 (9.7) | 61.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 62 | 119
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 47 | 56 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 62 | 119

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Urinary Retention
Description: Failed voiding trial upon removal of catheter
Time Frame: Within 72 hours of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tamsulosin
Number analyzed (Participants) | 62 | 57
Participants | 16 | 5

2. Secondary Outcome: International Prostate Symptom Score
Description: Total and subscale scores reported. Total score range 0-35, with 0 being less symptomatic and 35 being more symptomatic. Total score is sum of individual questions. Seven subgroups address incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining, nocturia. Each subgroup is scored 0-5 with 5 being most symptomatic. The last question is independent, rates quality of life from 0 (best) to 6 (worst)
Time Frame: Within 1 week of surgery
Measure: Median (Inter-Quartile Range); unit: Points
Arm/Group | Placebo | Tamsulosin
Number analyzed (Participants) | 37 | 35
Points | 6 [3 to 12.5] | 7 [3 to 11]

3. Secondary Outcome: Postoperative Urinary Tract Infection
Description: Treated for urinary tract infection with antibiotics or urinalysis or urine culture suggests infection.
Time Frame: Within 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tamsulosin
Number analyzed (Participants) | 62 | 57
Participants | 6 | 4

4. Secondary Outcome: Sent Home With Catheterization
Description: Urinary retention that required homegoing catheterization
Time Frame: within 6 weeks of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tamsulosin
Number analyzed (Participants) | 62 | 57
Participants | 7 | 5

ADVERSE EVENTS:
Time Frame: Three days prior to surgery through five days after surgery (10d total)
Arm/Group | Placebo | Tamsulosin
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/57
Serious Adverse Events (participants affected / at risk) | 2/62 | 1/57
Other Adverse Events (participants affected / at risk) | 3/62 | 3/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Tamsulosin (N=57)
Development of atrial fibrillation (Cardiac disorders) | 0 | 1 — Postoperative
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Postoperative
Congestive heart failure (Cardiac disorders) | 1 | 0 — Postoperative
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Tamsulosin (N=57)
Dizziness/lightheadedness (Nervous system disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03524339/Prot_SAP_000.pdf